CLINICAL TRIAL: NCT04247698
Title: Prognostic Value of Hemodynamic Forces at Rest and Stress Compared to Adenosine and Dobutamine Stress Cardiac Magnetic Resonance
Brief Title: Hemodynamic Forces at Rest and Stress vs. Adenosine and Dobutamine Stress Cardiac Magnetic Resonance
Acronym: CMR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayat Aboutaleb Abdellah Abdelgalil, Assistant lecturer, Assiut University
Other Study IDs: HDF
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stress perfusion CMR has recently considered as one of the methods of choice for establishing the diagnosis of CAD based on its high diagnostic accuracy, lack of ionizing radiation as well as its ability to simultaneously assess the cardiac function, myocardial perfusion, and viability, however, there are some concerns on its suitability for assessment of myocardial perfusion in patients after coronary artery bypass graft surgery who suffer from recurrent angina. The study of hemodynamic forces offers a promising tool for further understanding of the interplay between the myocardium and blood as well as the mechanisms of cardiac filling. This work represents a retrospective follow up study of CMR data, available on CMR-database, from 112 patients with previous coronary artery bypass grafting (CABG) performed around 10 years before the initial CMR examination. The study subjects underwent stress CMR testing; using both stressors; dobutamine and adenosine (done on two separate occasions). Injection of gadolinium contrast medium for late gadolinium enhancement was done with adenosine stress testing for late gadolinium enhancement (LGE). Offline analysis of these data will be done with the use of dedicated software for assessment for myocardial ischemia together with quantitative measurements of the hemodynamic forces with the help of dedicated software (QStrain version 1.3.0.79; Medis, Leiden, the Netherlands).

DETAILED DESCRIPTION:
In total 112 patients who underwent coronary artery bypass surgery (CABG) subjected to stress CMR examination on two separate occasions with both stressors; dobutamine and adenosine for assessment of myocardial ischemia as result of typical /atypical angina pectoris. The results from dobutamine (namely, detection of wall motion abnormalities) and adenosine stress CMR (namely, detection of perfusion abnormalities) will be compared with the values obtained from the measures of the hemodynamic forces of the LV (i.e., changes in the intraventricular pressures during systole and diastole). The dimensionless root mean square (FRMS) is computed over the entire heartbeat as a measure of the overall force amplitude. In addition, LV global longitudinal strain (GLS) and LV global circumferential strain (GCS) will be measured using a CMR feature tracking techniques. The expected results are as follows: Dobutamine wall motion analysis in combination with perfusion imaging has the highest diagnostic accuracy for the detection of ischemia in patients after bypass surgery and outperforms pure dobutamine wall motion or perfusion analysis and adenosine perfusion. Whereas, perfusion imaging with both stressors reflects the extent of ischemia more precisely than wall motion analysis. Nevertheless, assessment of hemodynamic forces adds to the diagnostic accuracy as well as the prognostic value of stress CMR in post-CABG patients, in whom stress testing with either or both stressors might fail to precisely define myocardial ischemia or reflect an associated subtle cardiac dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established CAD and underwent coronary artery bypass graft surgery (CABG) performed around 10 years before the initial CMR examination. Who presented to CMR examination because of recurrent typical/ atypical angina.

Exclusion Criteria:

* All patients that were not able to withstand the condition of CMR examination
* Patients who had contraindications to the stressor agents used in stress CMR were not included in the analysis (i.e. bronchial asthma, high degree heart-block)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population are known to have coronary artery disease and underwent revascularization therapy via bypass surgery around 10 years before the initial CMR examination. Those presented with manifestations of recurrent post-CABG angina, with either typical or atypical presentation. Each patient had two CMR examinations on two occasions using both dobutamine and adenosine stress agents.
Sampling Method: Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of hard and soft cardiac events and their relation to initial positive or negative Stress-CMR-test. | 1 year
  Hard cardiac outcomes are defined defined as deaths that are attributed to coronary artery disease, and non-fatal myocardial infarction. While soft events are defined as angina, or repeat revascularization for progressive coronary artery disease.

SECONDARY OUTCOMES:
Definition of the prognostic value of vasodilator stress and inotropic stress-CMR in patients with chronic CAD and a history of CABG. | 1 year
  The capability of both stressors to detect precisely the presence recurrent ischaemia in patients with CAD on both CMR examinations
Evaluation of the diagnostic accuracy of hemodynamic forces and assessment of the relationship to inducible wall motion abnormalities and perfusion defects. | 1 year
  The power of how much the analysis of hemodynamic forces in comparison to adenosine and dobutamine to precisely detect ischaemic changes in either positive and negative stress CMR in such patients

CONTACTS AND LOCATIONS:
Overall Officials: Amr Youssef, MD, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No